CLINICAL TRIAL: NCT04308616
Title: Utility of Squamous Cell Carcinoma Antigen (SCCA) in Psoriasis
Acronym: SCCAPSO
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI19/SCCAPSO; 2020-A00105-34 (Other: IdRCB)
Record Dates: First submitted 2020-03-05; First posted 2020-03-16 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Psoriasis
Keywords: Psoriasis; Squamous Cell Carcinoma Antigen; SCCA; Biomarker
MeSH Terms: conditions — Psoriasis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Psoriasis: Patients with psoriasis
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — Blood samples

SUMMARY:
Squamous Cell Carcinoma Antigen (SCCA) contributes to the pathogenesis of psoriasis by inhibiting cell apoptosis, exacerbating epidermal hyperplasia and skin inflammation. Three studies have shown a correlation between blood levels of SCCA and the severity of psoriasis.

Clinical scores of psoriasis severity are used in consultation to guide treatment of the disease (initiation of systemic therapy, dose escalation) but they suffer from several pitfalls: lack of inter- and intra-observer reproducibility, consumption of medical time.

A readily available, inexpensive (24 euros) blood marker could be an interesting alternative to these clinical scores.

DETAILED DESCRIPTION:
Squamous Cell Carcinoma Antigen (SCCA) contributes to the pathogenesis of psoriasis by inhibiting cell apoptosis, exacerbating epidermal hyperplasia and skin inflammation. Three studies have shown a correlation between blood levels of SCCA and the severity of psoriasis.

Clinical scores of psoriasis severity are used in consultation to guide treatment of the disease (initiation of systemic therapy, dose escalation). The PASI (Psoriasis Assessment Severity Index, minimum score 0, maximum 72) is the most widely used. It suffers from several pitfalls: lack of inter- and intra-observer reproducibility, consumption of medical time. This PASI score was "unavoidable" in the international clinical studies used to obtain marketing authorisation for medicines. The PGA (Physician global assessment) is simpler and less time-consuming, ranging from 0 to 4, but is not very discriminating. More recently, a "Simplified Psoriasis Index" (proSPI) health professional score has been developed, which correlates well with PASI for the severity component of psoriasis and with quality of life for the psychological component of the disease. It is less time-consuming to establish than PASI, but suffers like all clinical scores from a problem of inter- and intra-observer reproducibility.

A readily available, inexpensive (24 euros) blood marker could be an interesting alternative to these clinical scores.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patient with skin psoriasis (new and untreated or being treated, flare-up or stable, possibly bleached)
* Requiring a blood sample for disease or treatment monitoring

Exclusion Criteria:

* History of invasive mucosal squamous cell carcinoma, or squamous cell carcinoma of the skin with lymph node or visceral recurrence.
* Patient under guardianship or curatorship
* Opposition to participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with psoriasis
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
SCCA blood concentration | Baseline, 3 months and 6 months
  SCCA blood concentration will be measured at each visit

SECONDARY OUTCOMES:
Assess correlations between SCCA blood concentration and proSPI severity score | Baseline, 3 months and 6 months
  proSPI severity score (0-50) will be evaluated at each visit
Assess correlations between SCCA blood concentration and proSPI psychosocial score | Baseline, 3 months and 6 months
  proSPI psychosocial score (0-10) will be evaluated at each visit
Assess correlations between SCCA blood concentration and proSPI treatment score | Baseline, 3 months and 6 months
  proSPI treatment score (0-10) will be evaluated at each visit
Assess correlations between SCCA blood concentration and C reactive protein (CRP) | Baseline, 3 months and 6 months
  CRP will be measured at each visit
Assess correlations between SCCA blood concentration and neutrophil/lymphocyte ratio | Baseline, 3 months and 6 months
  neutrophil/lymphocyte ratio will be measured at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Laurent MACHET, MD-PhD, Principal Investigator — University Hospital, Tours
Locations (1):
- Dermatology Service, University Hospital, Tours, Tours, France